CLINICAL TRIAL: NCT02216656
Title: A Randomized, Double-blind, Parallel-group, Dose-finding Study of KHK7580 for Secondary Hyperparathyroidism Patients Receiving Hemodialysis
Brief Title: Phase 2 Study of KHK7580
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7580-005
Record Dates: First submitted 2014-08-11; First posted 2014-08-15 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Plascebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KHK7580 low dose (Experimental)
  Interventions: Drug: KHK7580 low dose
- KHK7580 middle dose (Experimental)
  Interventions: Drug: KHK7580 middle dose
- KHK7580 high dose (Experimental)
  Interventions: Drug: KHK7580 high dose
- KRN1493 (Active Comparator)
  Interventions: Drug: KRN1493

INTERVENTIONS:
Drug: Placebo — Oral administration
  Arms: Plascebo
Drug: KHK7580 low dose — Oral administration
  Arms: KHK7580 low dose
Drug: KHK7580 middle dose — Oral administration
  Arms: KHK7580 middle dose
Drug: KHK7580 high dose — Oral administration
  Arms: KHK7580 high dose
Drug: KRN1493 — Oral administration
  Other Names: cinacalcet
  Arms: KRN1493

SUMMARY:
This randomized, placebo-controlled, double-blind (included open arm of KRN1493 (cinacalcet)), parallel-group, multi-center study is designed to evaluate efficacy and safety in cohorts comprising KHK7580, its placebo and KRN1493 (cinacalcet) orally administered for three weeks for secondary hyperparathyroidism patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have voluntarily consented to participate in this study
* Subjects with stable chronic renal disease receiving hemodialysis 3 times weekly for at least 12 weeks before screening
* Subjects with an intact Parathyroid hormone of >= 240 pg/mL at screening

Exclusion Criteria:

* Subjects with primary hyperparathyroidism
* Subjects who have received cinacalcet hydrochloride within 2 weeks before screening
* Subjects whose dose or dosing regimen of an active vitamin D drug or its derivative, phosphate binders, or calcium preparation has been changed or started within 2 weeks before screening.
* Subjects who have underwent parathyroidectomy and/or parathyroid intervention within 24 weeks before screening.
* Subjects with uncontrolled hypertension and/or diabetes
* Subjects with severe heart disease.
* Subjects with severe hepatic dysfunction.
* Subjects who have received any other investigational drug within 12 weeks before screening
* Other subjects unfit for participation in this study in the judgment of the investigator or sub investigator.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The percent changes in intact Parathyroid hormone levels from baseline | Up to 3 weeks
  Percent changes in intact Parathyroid hormone levels from baseline to end of administration period

SECONDARY OUTCOMES:
Change from baseline in intact Parathyroid hormone , whole Parathyroid hormone, corrected serum Ca, ionized Ca, serum phosphorus, intact fibroblast growth factor 23 and corrected serum Ca X serum phosphorus. | Up to 3 weeks
  Change from baseline in intact Parathyroid hormone , whole Parathyroid hormone, corrected serum Ca, ionized Ca, serum phosphorus, intact fibroblast growth factor 23 and corrected serum Ca X serum phosphorus from baseline to end of administrations period.
Safety | Up to 3 weeks
  1. Number and types of adverse events
  2. laboratory tests
  3. vital signs
  4. 12-lead electrocardiogram
  5. ophthalmological examination

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Tokyo, Japan